CLINICAL TRIAL: NCT01021020
Title: Randomized, 3-Way Crossover Bioequivalence Study of Single Dose Colchicine Tablets and Effect of Food
Brief Title: Bioequivalence Study of Colchicine Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Vice President, Branded Products and Medical Affairs, Mutual Pharmaceutical Company, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MPC-004-07-1001
Record Dates: First submitted 2009-08-12; First posted 2009-11-26 (Estimated); Results first posted 2009-11-26 (Estimated); Last update posted 2009-12-09 (Estimated); Status verified 2009-12

CONDITIONS: Healthy
Keywords: bioequivalence; fasting; fed; healthy
MeSH Terms: conditions — Fasting; Lecithin Cholesterol Acyltransferase Deficiency | interventions — Colchicine; Probenecid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Colchicine (fasted)
  Interventions: Drug: Colchicine
- 2 (Experimental): Colchicine (fed)
  Interventions: Drug: Colchicine
- 3 (Active Comparator): Colchicine/Probenecid (fasted)
  Interventions: Drug: Colchicine/Probenecid

INTERVENTIONS:
Drug: Colchicine — 0.6mg tablet administered after a fast of at least 10 hours
  Other Names: COLCRYS TM
  Arms: 1
Drug: Colchicine — 0.6mg tablet administered after a standardized high-fat, high-calorie breakfast
  Other Names: COLCRYS TM
  Arms: 2
Drug: Colchicine/Probenecid — 0.5mg/500mg tablet administered after a fast of at least 10 hours
  Arms: 3

SUMMARY:
This randomized, single dose, three-way crossover study will evaluate the bioequivalence of two formulations of colchicine, the test product (colchicine 0.6mg Mutual) and a marketed combination product (colchicine 0.5 mg with probenecid 500 mg), administered under fasting conditions. It will also determine the bioavailability following a standard high-fat meal and evaluate the safety and tolerability of the test product.

DETAILED DESCRIPTION:
This randomized, single dose, three-way crossover study will evaluate the bioequivalence of two formulations of colchicine, the test product (colchicine 0.6mg Mutual) and a marketed combination product (colchicine 0.5mg with probenecid 500mg), administered under fasting conditions. It will also determine the bioavailability of the test product following a standard high-fat meal and evaluate the safety and tolerability of the test product. Twenty-eight healthy, non-smoking, non-obese (BMI 81-30 kg/m2 and BW ≥110 lbs), 18-45 year old, male and female volunteers will be randomly assigned in a crossover fashion to receive one of three dosing regimens in sequence with washout periods of at least 14 days between dosing periods. After a fast of at least 10 hours, subjects will receive either, one tablet of colchicine 0.6 mg, one tablet of colchicine 0.6 mg after a standardized high-fat,high-calorie breakfast or 0.5mg/500mg colchicine/probenecid. All doses will be given with 240mL of room temperature water. Patients will be confined for at least 15 hours before and 24 hours after each dose with daily outpatient visits over the following 3 days. Blood will be drawn at times sufficient to adequately define the concentration time curves for each dosing regimen, which will be compared to assess the bioequivalence of the reference and test products and the effect of food on the test product. Subjects will also be monitored for adverse events throughout this same period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers, male and female, 18 to 45 years of age, inclusive, with BMI between 18-30 kg/m2, inclusive, and weighing at least 110 pounds.
* Female volunteers must be postmenopausal, surgically sterile, or must commit to abstain from heterosexual contact or to use two methods of reliable birth control.

Exclusion Criteria:

* Subjects who report receiving any investigational drug within 28 days prior to initiation of dosing.
* Subjects who report presence or history of significant cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, neurologic, or psychiatric disease.
* Subjects with clinical lab results outside accepted reference range, or reactive screen for hepatitis B surface antigen, hepatitis C antibody, or HIV antibody.
* Subjects who report a history of allergies to colchicine or related drugs, or history of other clinically significant allergies including drug allergies.
* Subjects who report a clinically significant illness during the 4 weeks prior to initiation of dosing.
* Subjects who report a history of drug or alcohol addiction or abuse within the past year, or who demonstrate a positive drug abuse screen.
* Subjects who currently use or have used tobacco products within 6 months prior to dose administration.
* Subjects who report donating greater than 150 ml of blood within 28 days or donating plasma within 14 days prior to initiation of dosing.
* Subjects who have a positive pregnancy screen, or are currently pregnant or breastfeeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2007-09; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony R Godfrey, Pharm.D., Principal Investigator — PRACS Institute, Ltd.
Locations (1):
- PRACS Institute, Ltd. - Cetero Research, Fargo, North Dakota, United States

REFERENCES:
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html
- See also: Daily Med - Posting of Recently Submitted Labeling to the FDA — http://dailymed.nlm.nih.gov/dailymed/about.cfm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-eight (28) healthy, non-smoking, adult male and female volunteers, consisting of university students and members of the community at large, were to be enrolled.
Pre-assignment Details: 75 subjects screened, 47 were screen failures
Groups:
- Colchicine (Fasted),Colchicine (Fed),Colchicine/Probenecid: All subjects received each of the three study treatments in a randomly assigned sequence of dosing periods. On the morning of Days 1, 15, and 29, each subject received one of the following three treatments: 1) one tablet of colchicine 0.6 mg after an overnight fast of at least 13.5 hours, 2) one tablet of colchicine 0.6 mg after a high-fat breakfast, or 3) one tablet of colchicine 0.5 mg/ probenecid 500 mg following an overnight fast of at least 13.5 hours.
Period: Period I
Arm/Group | Colchicine (Fasted),Colchicine (Fed),Colchicine/Probenecid
Started | 28
Completed | 26 (Colchicine(fasted)-subject took Claritin-D 12hour.Colchicine(fed)arm-subject had schedule conflict.)
Not Completed | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1
Period: 14 Day Washout Period A
Arm/Group | Colchicine (Fasted),Colchicine (Fed),Colchicine/Probenecid
Started | 26
Completed | 25 (Colchicine/Probenecid-medical investigator dropped due to abnormal check-in lab results.)
Not Completed | 1
Not completed — Physician Decision | 1
Period: Period II
Arm/Group | Colchicine (Fasted),Colchicine (Fed),Colchicine/Probenecid
Started | 25
Completed | 25
Not Completed | 0
Period: 14 Day Washout Period B
Arm/Group | Colchicine (Fasted),Colchicine (Fed),Colchicine/Probenecid
Started | 25
Completed | 25
Not Completed | 0
Period: Period III
Arm/Group | Colchicine (Fasted),Colchicine (Fed),Colchicine/Probenecid
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Colchicine(Fasted),Colchicine(Fed),Colchicine/Probenecid: All subjects received all study treatments in a randomly assigned sequence of dosing periods. On the morning of Days 1, 15, and 29, each subject received one of the following three treatments: 1) one tablet of colchicine 0.6 mg after an overnight fast of at least 13.5 hours, 2) one tablet of colchicine 0.6 mg after a high-fat breakfast, or 3) one tablet of colchicine 0.5 mg/ probenecid 500 mg following an overnight fast of at least 13.5 hours.
Arm/Group | Colchicine(Fasted),Colchicine(Fed),Colchicine/Probenecid
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants] — age range: >=18 and <=45 years old
  Participants
    <=18 years | 0
    Between 18 and 65 years | 28
    >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 23.7 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 24
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Maximal Plasma Concentration (Cmax)
Description: The maximum or peak concentration that colchicine reaches in the plasma.
Time Frame: serial pharmacokinetic blood samples collected pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72 and 96 hours post-dose
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Colchicine 0.6 mg (Fasted): Subjects received one tablet of colchicine 0.6 mg after an overnight fast.
- Colchicine (High-fat Meal): Subjects received one tablet of colchicine 0.6 mg after a high-fat breakfast.
- Colchicine 0.5 mg/ Probenecid 500 mg (Fasted): Subjects received one tablet of colchicine 0.5 mg/ probenecid 500 mg following an overnight fast.
Arm/Group | Colchicine 0.6 mg (Fasted) | Colchicine (High-fat Meal) | Colchicine 0.5 mg/ Probenecid 500 mg (Fasted)
Number analyzed (Participants) | 25 | 25 | 25
pg/mL | 2,503.04 (722.05) | 2,496.88 (695.09) | 1,706.03 (560.73)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the plasma concentration versus time curve, from time 0 to the time of the last measurable colchicine concentration (t), as calculated by the linear trapezoidal rule.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg-hr/mL
Groups:
- Colchicine 0.6 mg (Fasting): Subjects received one tablet of colchicine 0.6 mg after an overnight fast.
- Colchicine 0.6 mg (High-fat Meal): Subjects received one tablet of colchicine 0.6 mg after a high-fat meal.
- Colchicine 0.5 mg/ Probenecid 500 mg (Fasting): Subjects received one tablet of colchicine 0.5 mg/ probenecid 500 mg following an overnight fast
Arm/Group | Colchicine 0.6 mg (Fasting) | Colchicine 0.6 mg (High-fat Meal) | Colchicine 0.5 mg/ Probenecid 500 mg (Fasting)
Number analyzed (Participants) | 25 | 25 | 25
pg-hr/mL | 12,588.61 (6,120.73) | 10,490.95 (4,025.80) | 8,090.05 (6,111.99)

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 Extrapolated to Infinity [AUC(0-∞)]
Description: The area under the plasma concentration versus time curve from time 0 to infinity. AUC(0-∞) was calculated as the sum of AUC(0-t) plus the ratio of the last measurable colchicine plasma concentration to the elimination rate constant.
Time Frame: as for outcome 1
Population: Colchicine(fasted)-could not be determined for Subject 25. Colchicine(high-fat meal)-could not be determined for Subjects 22,25, and 28. Colchicine/Probenecid(fasted)-could not be determined for Subject 25.
Measure: Mean (Standard Deviation); unit: pg-hr/mL
Groups:
- Colchicine 0.6 mg (High-fat Meal): Subjects received one tablet of colchicine 0.6 mg after a high-fat breakfast.
Arm/Group | Colchicine 0.6 mg (Fasted) | Colchicine 0.6 mg (High-fat Meal) | Colchicine 0.5 mg/ Probenecid 500 mg (Fasted)
Number analyzed (Participants) | 24 | 22 | 24
pg-hr/mL | 14,112.52 (5,595.40) | 11,404.09 (2,895.68) | 8,481.41 (2,829.75)

ADVERSE EVENTS:
Description: 28 subjects were enrolled in this study. Several subjects dropped out of the study prior to receiving all interventions. 26 subjects were administered colchicine 0.6 mg tablets (fasted). 27 subjects were administered colchicine 0.6 mg tablets(fed). 27 subjects were co-administered colchicine 0.5 mg/probenecid 500 mg tabs (fasted).
Groups:
- Colchicine 0.6 mg (Fasted): Subjects received one tablet of colchicine 0.6mg after an overnight fast of at least 13.5 hours.
- Colchicine 0.6 mg (Fed): Subjects received one tablet of colchicine 0.6 mg after a high-fat meal.
- Colchicine 0.5 mg/Probenecid 500 mg (Fasted): Subjects received one tablet of colchicine 0.5 mg/ probenecid 500 mg after an overnight fast of at least 13.5 hours.
Arm/Group | Colchicine 0.6 mg (Fasted) | Colchicine 0.6 mg (Fed) | Colchicine 0.5 mg/Probenecid 500 mg (Fasted)
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 5/26 | 3/27 | 4/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colchicine 0.6 mg (Fasted) (N=26) | Colchicine 0.6 mg (Fed) (N=27) | Colchicine 0.5 mg/Probenecid 500 mg (Fasted) (N=27)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
stomach discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
paresthesia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2)
headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
sinus headache (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days